CLINICAL TRIAL: NCT05112237
Title: A Prospective and Retrospective Registry and Biomarker Study to Evaluate the Natural History of Pediatric Patients With Cardiomyopathy Due to MYBPC3 Mutations
Brief Title: Natural History Study in Pediatric Patients With MYBPC3 Mutation-associated Cardiomyopathy
Acronym: MyCLIMB
Status: Recruiting | Type: Observational
Sponsor: Tenaya Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: TN-201-0003
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Cardiomyopathy
Keywords: Genetic Cardiomyopathy; Pediatric; MYBPC3; Hypertrophic Cardiomyopathy (HCM); Dilated Cardiomyopathy; Restrictive Cardiomyopathy; Non-Compaction cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies; Cardiomyopathy, Hypertrophic; Cardiomyopathy, Dilated; Cardiomyopathy, Restrictive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: All patients who meet the eligibility criteria will be eligible for retrospective chart review.
- Prospective: 100 patients meeting the eligibility criteria will be followed for 5 years, in addition to a retrospective chart review. Assessments will be completed as part of a participant's regular schedule of physician visits, no additional visits will be required. Aside from a simple annual blood draw, assessments are non-invasive, including a Quality of Life questionnaire.

SUMMARY:
The objective of this study is to collect information on patients with cardiomyopathy (CM) due to mutations in the MYBPC3 gene, to evaluate their disease course, burden of illness, risk factors for this disease, and the quality of life (QoL). This study will also collect information on treatments, procedures and outcome in infants and children up to 18 yrs who have this mutation.

ELIGIBILITY:
Retrospective

Inclusion Criteria:

* Data is available for patient <18 years of age. Patients must be <18 years of age at enrollment or at time of death.
* Documented results of genotyping showing the presence of at least one pathogenic or likely pathogenic MYBPC3 mutation (heterozygous, homozygous, or compound heterozygous).

Exclusion Criteria:

* Patient received cardiac transplantation or died >10 years before study initiation. For homozygous or biallelic infants, data may be collected beyond this 10-year period.

Prospective

Inclusion Criteria:

For Infants:

* Infants who are homozygous or compound heterozygous for the known pathogenic truncating MYBPC3 mutations are eligible.

For all other participants:

* Age <18 at entry into the prospective study.
* Documented results of genotyping identifying at least one pathogenic or likely pathogenic MYBPC3 mutation (heterozygous, homozygous, or compound heterozygous).
* Diagnosis of Cardiomyopathy (CM): HCM, DCM, RCM, mixed CM, or LVNC.

Exclusion Criteria:

* Concurrent participation in an interventional clinical trial unless approved by the sponsor.
* Severe noncardiac disease anticipated to significantly reduce life expectancy.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients under the age of 18 years (at enrollment) with cardiomyopathy (CM) and pathogenic or likely pathogenic MYBPC3 genetic mutation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
To characterize the disease course and natural history in participants with pathogenic or likely pathogenic MYBPC3 mutations with a specific focus on cardiac events and measurement | 5 years for prospective group, n/a for retrospective group

CONTACTS AND LOCATIONS:
Locations (29):
- United States (21):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California Davis Health, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of Colorado Hospital - Anschutz Medical Campus, Aurora, Colorado
  - Nemours Alfred I. Dupont Hospital for Children, Wilmington, Delaware
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Children's Mercy Hospital Kansas, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Cohen Children's Medical Center, Lake Success, New York
  - Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - DDC Clinic Center for Special Needs Children, Middlefield, Ohio
  - Cardiology Care for Children, Lancaster, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - The Hospital for Sick Children, Toronto, Ontario
- Spain (3):
  - Hospital Sant Joan de Déu Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Alvaro Cunqueiro - Clinico Universitario Vigo, Vigo
- United Kingdom (3):
  - NHS Greater Glasgow and Clyde, Glasgow
  - Royal Brompton & Harefield NHS Foundation Trust, London
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No